CLINICAL TRIAL: NCT05762445
Title: A Patient-Driven Registry for Exocrine Pancreatic Insufficiency Due to Chronic Pancreatitis
Brief Title: PAtient-CenTric Chronic Pancreatitis Registry (PACT-CP)
Acronym: PACT-CP
Status: Completed | Type: Observational
Sponsor: CorEvitas (Network)
Collaborators: Nestle Health Science (Industry)
Responsible Party: Sponsor
Other Study IDs: NES-EPI-100
Record Dates: First submitted 2022-01-20; First posted 2023-03-09 (Actual); Last update posted 2026-01-22 (Actual); Status verified 2026-01

CONDITIONS: Chronic Pancreatitis
MeSH Terms: conditions — Pancreatitis, Chronic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
The main objective of this study is to generate real-world evidence reflecting the experience of individuals with exocrine pancreatic insufficiency (EPI) due to chronic pancreatitis (CP). Efforts will be directed toward understanding the unmet need and therapeutic burden to identify the most critical factors that influence treatment choices/prescribing patterns, quality of life, and healthcare utilization outcomes in standard of care for individuals with EPI due to CP.

DETAILED DESCRIPTION:
Study participants will be followed prospectively, and data from study participants will be collected at 3-month intervals via Electronic Data Capture (EDC) portal. Investigators will complete assessments approximately every 6 months at the time of routine clinical encounters. Adverse Events (AEs) will be collected as part of the study data collection forms. Serious Adverse Events (SAEs) are to be reported within 24 hours (1 business day) of awareness, whether or not the site learns of the event at the time of a registry follow-up visit.

ELIGIBILITY:
Inclusion Criteria:

To be eligible for enrollment, a study participant must meet the inclusion criteria below:

1. At least 18 years of age (or age of majority)
2. Willing to provide consent to participate
3. Meet one (1) of the following at the time of enrollment:

   1. Diagnosis of chronic pancreatitis (CP)
   2. Diagnosis of recurrent acute pancreatitis (RAP)
4. Suspected or confirmed diagnosis of EPI made by a healthcare provider
5. On Pancreatic Enzyme Replacement Therapy (PERT), either prior to the Enrollment Visit or newly prescribed at the time of the Enrollment Visit.

To be eligible for enrollment into the registry, a study participant must not have any of the criteria below:

1. Currently participating in or planning to participate in a double-blind randomized trial and/or open-label Phase 3b/4 on CP or EPI
2. Diagnosed with any of the following conditions at the time of enrollment:

   1. Cystic fibrosis
   2. Fibrosing colonopathy
   3. A history of or current diagnosis of pancreatic cancer, main duct papillary mucinous neoplasms (IPMNs), and other pancreatic malignancies
   4. Allergy to pork or other porcine pancreatic enzyme products (PEPs)
   5. Any condition that would, in the investigator's opinion, limit the individual's ability to complete the study.

      -

      Exclusion Criteria:

      -

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This is a prospective, non-interventional study for individuals with EPI due to CP who are under the care of a gastroenterologist.
Sampling Method: Non-Probability Sample
Enrollment: 400 (Actual)
Dates: Start 2021-06-02 (Actual); Primary Completion 2025-08-31 (Actual); Study Completion 2025-08-31 (Actual)

PRIMARY OUTCOMES:
Main Objective of the Study | Up to 5 years
  The main objective of this study is real-world evidence reflecting the experience of individuals with exocrine pancreatic insufficiency (EPI) due to chronic pancreatitis (CP).
Creation of a Patient Cohort | Up to 5 years
  Create a cohort of well-characterized patients with EPI due to CP research.
Disease History and Progression Data at Initial Visit | At Initial Visit
  Collect clinical data to characterize both the EPI due to CP disease history and disease progression at the initial visit.
Progression Data (Every 3 months after Initial Visit) | Every 3 months after Initial Visit up to 5 years
  Collect clinical data to characterize EPI due to CP disease progression every 3 months after the initial visit through a patient reported outcome (PRO).
Progression Data (Every 6 months after Initial Visit) | Every 6 months after Initial Visit up to 5 years
  Collect clinical data to characterize EPI due to CP disease progression every 6 months after the initial visit alongside the physician at the site.
Clinical Care Practice Data at Initial Visit | At Initial Visit
  Collect data on clinical care practices for participants with EPI to better understand the impact on outcomes at the initial visit.
Clinical Care Practice Data (Every 3 months after Initial Visit) | Every 3 months after Initial Visit up to 5 years
  Collect data on clinical care practices for participants with EPI to better understand the impact on outcomes every 3 months after the initial visit through a patient reported outcome (PRO).
Clinical Care Practice Data (Every 6 months after Initial Visit) | Every 6 months after Initial Visit up to 5 years
  Collect data on clinical care practices for participants with EPI to better understand the impact on outcomes every 6 months after the initial visit alongside the physician at the site.
Treatment Compliance Data at Initial Visit | At Initial Visit
  Collect data on treatment compliance that may impact the EPI due to CP disease experience and/or outcome at the initial visit.
Treatment Compliance Data (Every 3 months after Initial Visit) | Every 3 months after Initial Visit up to 5 years
  Collect data on treatment compliance that may impact the EPI due to CP disease experience and/or outcome every 3 months after the initial visit through a patient reported outcome (PRO).
Treatment Compliance Data (Every 6 months after Initial Visit) | Every 6 months after Initial Visit up to 5 years
  Collect data on treatment compliance that may impact the EPI due to CP disease experience and/or outcome every 6 months after the initial visit alongside the physician at the site.
Baseline Data | At Initial Visit
  Collect baseline data of participants with EPI due to CP at the initial visit.
PRO Data | Every 3 months after Initial Visit up to 5 years
  Collect longitudinal participant-reported outcome (PRO) data every 3 months after Initial Visit.
Impact and Burden of EPI due to CP Data at Initial Visit | At Initial Visit
  Gather data on healthcare utilization to be combined with clinical data to generate evidence for the impact and burden of EPI due to CP in this cohort on the healthcare system at the initial visit.
Impact and Burden of EPI due to CP (Every 3 months after Initial Visit) | Every 3 months after Initial Visit up to 5 years
  Gather data on healthcare utilization to be combined with clinical data to generate evidence for the impact and burden of EPI due to CP in this cohort on the healthcare system every 3 months after the initial visit through a patient reported outcome (PRO).
Impact and Burden of EPI due to CP (Every 6 months after Initial Visit) | Every 6 months after Initial Visit up to 5 years
  Gather data on healthcare utilization to be combined with clinical data to generate evidence for the impact and burden of EPI due to CP in this cohort on the healthcare system every 6 months after the initial visit alongside the physician at the site.

CONTACTS AND LOCATIONS:
Overall Officials: David Whitcomb, MD, PhD, Study Chair — Director, University of Pittsburgh Medical Center; Jodie Barkin, MD, Study Chair — University of Miami, Division of Gastroenterology; Samer Al-Kaade, MD, Study Chair — Mercy Clinic Gastroenterology; Yasmin Hernandez-Barco, MD, Study Chair — Harvard School of Medicine, Division of Gastroenterology and Hepatology; Rahul Pannala, MD, Study Chair — Mayo Clinic College of Medicine and Science
Locations (1):
- CorEvitas, Waltham, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (3):
  • Study Protocol (2021-04-13): https://cdn.clinicaltrials.gov/large-docs/45/NCT05762445/Prot_000.pdf
  • Statistical Analysis Plan (2021-07-14): https://cdn.clinicaltrials.gov/large-docs/45/NCT05762445/SAP_001.pdf
  • Informed Consent Form (2021-04-08): https://cdn.clinicaltrials.gov/large-docs/45/NCT05762445/ICF_002.pdf